CLINICAL TRIAL: NCT05881967
Title: Molecular Mechanism Study of Uterine Sarcoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shixuan Wang (Other)
Responsible Party: Sponsor-Investigator, Shixuan Wang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: IRB20221166
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Uterine Sarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uterine sarcoma: Participants were enrolled for the first treatment of uterine sarcoma or secondary operation for recurrence fo uterine sarcoma.
  Interventions: Diagnostic Test: Diagnostic biomarker
- Uterine fibroid: Participants were enrolled for surgery of uterine fibroids.
  Interventions: Diagnostic Test: Diagnostic biomarker

INTERVENTIONS:
Diagnostic Test: Diagnostic biomarker — Diagnostic gene for uterine sarcoma

SUMMARY:
The purpose of this project was to use multi-omics technology to screen the key factors for the occurrence and development of uterine sarcoma.

DETAILED DESCRIPTION:
Uterine sarcomas are rare mesenchymal neoplasms in the female genital system, accounting for about 1% of female reproductive tract malignancies and 3%~7% of uterine malignancies. Subtypes of uterine sarcoma are leiomyosarcoma, endometrial stromal sarcoma, and adenosarcoma. Uterine leiomyosarcoma is the most common uterine sarcoma, accounting for about 1% to 2% of all uterine malignancies.

Uterine sarcomas differ in histologic appearance and clinical behavior. The incidence of uterine sarcoma is low and the prognosis is poor. Its manifestations mainly include abnormal vaginal bleeding, abdominal pain and abdominal mass, but none of these symptoms are specific.

For uterine sarcoma, there are no diagnostic serum markers and imaging features and the diagnosis of uterine sarcoma still mainly depends on postoperative pathological results. However, with the development of omics technology, immunophenotypes and molecular characterization of uterine sarcomas have increasingly been utilized to improve diagnostic classification and prognostication in uterine sarcomas. Uterine leiomyosarcoma, the most common subtype of uterine sarcoma, does not have a single defining molecular abnormality.

This project intends to use multi-omics technology to screen the key factors for the occurrence, development, and malignant transformation of uterine sarcoma, especially uterine leiomyosarcoma, and to map the interaction network of cell signaling pathways. It provides key molecular markers for the early assessment of recurrence and malignant transformation of uterine myoma after conservative treatment, and provides a molecular mechanism basis for finding solutions to prevent the progression and malignant transformation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older;
2. Newly treated or recurenced uterine sarcoma.

Exclusion Criteria:

1. Diagnosis of other malignancies within the past 5 years;
2. history of pelvic or vaginal radiation therapy;
3. Known high-grade lesions of the cervix and endometrium.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 patients who met the requirements includ 200 uterine sarcomas, 200 uterine leiomyomas.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Susceptible gene in women with uterine sarcoma | baseline
  Analyze genetic susceptibility among women exhibiting disease manifestations of uterine sarcoma

CONTACTS AND LOCATIONS:
Locations (1):
- Yan Li, Wuhan, Hubei, China